CLINICAL TRIAL: NCT02164630
Title: Assessing the Efficacy of a Hope Intervention in Temporomandibular Disorder
Brief Title: Optimizing Resilience In Orofacial Pain and Nociception
Acronym: ORION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: American Pain Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB201400260
Record Dates: First submitted 2014-06-12; First posted 2014-06-16 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Temporomandibular Joint Disorder
Keywords: Temporomandibular Joint Disorder; TMD; Hope; Resilience; Cognitive Behavior Therapy
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hope Therapy (Experimental): Patients assigned to this arm will receive Hope Therapy in three individual intervention sessions. Intervention will be administered by an experienced therapist.Training focuses on effective goal setting and augmenting hopeful thinking.
  Interventions: Behavioral: Hope Therapy
- Pain Education (Other): Patients assigned to this arm will receive Pain Education in three individual intervention sessions. Intervention will be administered by an experienced therapist. Training will focus on understanding TMD-related pain and learning pain management techniques.
  Interventions: Other: Pain Education

INTERVENTIONS:
Behavioral: Hope Therapy — Hope therapy is designed to address key components of hope theory through augmentation of hopeful thinking and enhancement of goal-directed activities. Training focuses on effective goal setting, mobilization of internal resources to reach goals, identification of resilience factors to formulate hopeful thinking, and enhancing maintenance of future goal development.
  Arms: Hope Therapy
Other: Pain Education — Pain Education is aimed to increase understanding of TMD symptomatology and etiology, as well as provide general education on pain, lifestyle management, and effective pain communication methods.
  Arms: Pain Education

SUMMARY:
The purpose of this study is to examine the effects of a hope-based intervention on clinical and experimental pain in individuals with temporomandibular disorder (TMD). To examine the effectiveness of this intervention, a two-arm randomized trial will be conducted with 50 individuals, between the ages of 18 and 65, who have TMD.

DETAILED DESCRIPTION:
In recent years, there has been increasing interest in the contribution of positive psychological factors (e.g., optimism, pain acceptance, hope) to pain and pain-related coping. Although research supports the significance of these resilience factors in pain adaptation, psychological interventions based upon bolstering resilience have received far less attention. Emerging evidence supports the role of hope in psychosocial adjustment and enhancement of adaptive pain coping skills. Hope is considered to be a positive motivational state consisting of one's belief in their ability to generate routes to achieve goals (pathways) and initiation towards attaining these goals (agency). In the context of pain, increasing hope may promote augmentation of personal strengths to enhance development of meaningful goal pursuits and foster resilient outcomes. Enhancement of hopeful thinking and behavior may ultimately lead to the minimization of losses that are often associated with chronic pain. This experience may be also reflected physiologically, as increasing hope may confer biological benefits (e.g., decreased inflammation). Although hope-based interventions have been successfully applied in other clinical conditions (i.e., cancer), their utility in chronic pain disorders has not been examined.

To examine the effectiveness of this approach, a two-arm randomized trial will be conducted with individuals who have TMD. In Study Arm 1, participants will receive hope-based therapy. In Study Arm 2, participants will receive pain education. Participants will attend 5 sessions over a period of 5 weeks. Two of these sessions will involve quantitative sensory pain testing; three sessions will include delivery of the treatment intervention. Pain outcomes will be measured at pre- and post-treatment.

Aims:

1. Examine the degree to which state and trait levels of hope are predictive of clinical pain, disability, affective distress, and experimental pain.
2. Investigate the effects of a hope intervention, as compared to an education control group, on clinical and experimental pain in individuals with TMD.
3. Identify psychosocial (e.g., hope, optimism, positive affect, catastrophizing), biological (e.g., inflammatory, endogenous opioid, neuroendocrine), and psychophysical factors associated with positive treatment response (i.e., reduction of clinical pain).

ELIGIBILITY:
Inclusion Criteria:

* participants between the ages of 18 and 65
* meets Research Diagnostic Criteria for TMD
* duration of pain is at least 3 months
* pain at least 15 days in the past month
* pain rated moderate to severe in intensity

Exclusion Criteria:

* uncontrolled hypertension
* current heart disease including heart failure
* kidney failure or currently undergoing dialysis
* current neurological conditions that could affect protocol safety or validity
* facial trauma or orofacial surgery within the last 6 months
* currently in orthodontic treatment
* currently pregnant and/or nursing
* use of narcotic analgesics (i.e., opioids) on a daily basis
* a primary pain condition other than TMD

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in state hope on the 8-point Adult State Hope Scale at week 5 | Baseline, Week 5
  The Adult State Hope Scale is a 6-item inventory used to assess goal-directed thinking at a given moment in time.
Change from baseline in clinical pain on the 0-100 Numerical Rating Scale at week 5 | Baseline, Week 5
  0-100 Numerical Rating Scale used to assess clinical pain intensity.

SECONDARY OUTCOMES:
Change from baseline in inflammatory, endogenous opioid, and neuroendocrine markers at week 5 | Baseline, Week 5
  Measurement of interleukin 6 (IL-6), beta-endorphin, cortisol, and alpha-amylase.
Change from baseline in optimism on the 5-point Life Orientation Test - Revised (LOT-R) at week 5 | Baseline, Week 5
  The LOT-R is a 10-item measure assessing generalized positive outcome expectancies.
Change from baseline in positive and negative affect on the 5-point Positive and Negative Affect Schedule (PANAS) scale at week 5 | Baseline, Week 5
  The PANAS is a 20-item scale that assesses positive affect (PA) and negative affect (NA).
Change from baseline in pain catastrophizing on the 5-point Pain Catastrophizing Scale (PCS) at week 5 | Baseline, Week 5
  The PCS is a 13-item measure used to assess patient report of catastrophic thinking about pain
Change from baseline in sensory pain stimuli at week 5 | Baseline, Week 5
  Measurement of heat pain threshold, heat pain tolerance, pressure pain threshold, cold pain threshold, and cold pain tolerance. Threshold = when stimulus (in seconds) is first rated as "painful"; Tolerance = when stimulus (in seconds) is no longer able to be tolerated.

CONTACTS AND LOCATIONS:
Overall Officials: Emily J Bartley, Ph.D., Principal Investigator — University of Florida
Locations (1):
- University of Florida, Pain Research and Intervention Center of Excellence (PRICE), Gainesville, Florida, United States